CLINICAL TRIAL: NCT05884619
Title: Efficacy and Safety of Dual-target Deep Brain Stimulation for Treatment-resistant Alcohol Use Disorder: a Multi-center, Single Arm, Prospective, Open-label, Extendable Study.
Brief Title: Efficacy and Safety of Dual-target Deep Brain Stimulation for Treatment-resistant Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Shanghai Mental Health Center (Other); Huashan Hospital (Other); Shanghai 6th People's Hospital (Other); SceneRay Corporation, Limited (Industry)
Responsible Party: Principal Investigator, Wei Hao, Chief Physician, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR1182-AUD-I
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use Disorder; Deep Brain Stimulation
Keywords: Alcoholism; Alcohol Drinking; Drinking Behavior; Alcohol-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Drinking Behavior; Alcohol-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-target deep brain stimulation (Experimental): This is a single arm, prospective, open label clinical study, participants who fit inclusion and don't fit exclusion criteria, completed physical anti-addiction treatments and surgical implantation standard will start DBS system stimulation and adjust parameters after 10-14 days of implantation. Then after stimulation for 9-32 weeks, they will be evaluated for treatment efficacies. This study is extendable, with agreements from participants, long term efficacy and safety follow-up study will be performed after 32 weeks ± 7 days of following, once every 2-3 months.
  Interventions: Device: Dual-target deep brain stimulation

INTERVENTIONS:
Device: Dual-target deep brain stimulation — DBS electrodes will be implanted into the ALIC and the NAcc, electric stimulation of those areas are used to treat alcohol use disorder and to evaluate the efficacy and safety of DBS system.

SUMMARY:
This is a multi-center, single arm, prospective, open-label, extendable study for the efficacy and safety of dual-target deep brain stimulation for treatment-resistant alcohol use disorder.

DETAILED DESCRIPTION:
Total of 12 subjects from two centers ( Shanghai Mental Health Center and The Second Xiangya Hospital of Central South University ) who meet inclusion and don't meet exclusion criteria are recruited to undergo neurosurgical implantation of dual-target DBS in bilateral nucleus accumbens (NAcc) and anterior limb of internal capsule (ALIC) on Day 0. The DBS system will be turned on for stimulation and parameter adjustment will be conducted on day 10-14 after implantation. The efficacy and safety evaluation will be conducted in 9-32 weeks after implantation. The indicators on efficacy are heaving drinking rate, uncontrolled alcohol consumption days, maximum consecutive alcohol abstinent days. The indicators for safety are adverse events (AE) and device related AE, serious adverse events (SAE) and device related SAE, device deficiencies (DD) and device malfunction, physical examination and vital signs, laboratory examination, ECG, imaging examination, scale evaluation and early drop out ratio due to AE.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old, no limit on sex.
2. Meet The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for alcohol use diagnosis with more than 4 positive items.
3. Course of alcohol use disorder ≥ 3 years.
4. Had at least 3 failed quit drinking experiences (de-addiction treatment under medical conditions, quit drinking by oneself, quit drinking each time ≥ 1 week)
5. Patient and relatives agree to accept systemic treatment of this study and sign Informed Consent Form after study purpose, content, expected treatment and risk etc. are fully explained and understood.

Exclusion Criteria:

1. Patients with other serious mental disorders (e.g. schizophrenia spectrum, depression disorder, biphasic or related disorder, etc. )
2. Patients who have other substance (other than tobacco) use disorders.
3. During screening period, answered 'yes' on question 4 or 5 in suicide intention term from Columbia-Suicide Severity Rating Scale, or had significant suicidal ideations in the past 3 months, or patients who are considered by researchers to have suicide or violence risks.
4. Patients who have serious or unstable cardiovascular, respiratory, liver, kidney, hematological, endocrine, nervous system or other systemic diseases.
5. Patients who have implanted cochlear, pacemaker, cardiac defibrillator, single-sided or double-sided products of the same category, or the investigator evaluates patients have done surgeries within 6 months that can affect this study.
6. HIV positive patients.
7. Woman at pregnant or lactation period, or childbearing age woman test positive for human chorionic gonadotropin (HCG)/urine pregnancy check; or patients who can't take effective contraception measures during trial; or patients who plan to be/make pregnant 3 months after the trial starts.
8. Patients who are participating other pharmaceutical or medical device clinical trials or have participated one in the past 3 months.
9. Patients who are considered unsuitable by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Heavy drinking rate | 9-32 weeks of stimulation
  Calculation formula: 'major alcohol use' times / 56 (total observation times) * 100%; a) Marked as maximum days of 'Constant alcohol suspension' b) Note: i. Major alcohol use standard: Blow test positive and reported ≥ 5 standard cups daily over the past 3 days. 1 standard cup = 10g of pure alcohol.
Cumulated uncontrolled alcohol use days | 9-32 weeks of stimulation
  Total days of all uncontrolled alcohol use days throughout 24 weeks
  1. Definition: more than 3 times consecutive alcohol use (random draw) ≥ 5 standard cups
  2. One time uncontrolled alcohol use days: e.g. 3 times consecutive follow-up results ≥ 5 standard cups, fourth time < 5 standard cups, then uncontrolled alcohol use days is 3 * 3 = 9 days
  3. Cumulated uncontrolled alcohol use days: Total days of all uncontrolled alcohol use days throughout 24 weeks
Maximum consecutive alcohol abstinent days | 9-32 weeks of stimulation
  Constant alcohol suspension standard: Blow test negative and no alcohol use reported over past 3 days.
  Marked as maximum days of 'Constant alcohol suspension'

SECONDARY OUTCOMES:
Alcohol use volume | 9-32 weeks after stimulation
  change in monthly average alcohol use volume compared to baseline. (Record in every follow-up according to participants. Record alcohol type, amount and experience when drinking throughout 9-32 weeks after stimulation. Increased value implies worse result and reduce of alcohol use volume indicates improvement.
Cumulated alcohol abstinent days | 9-32 weeks of stimulation.
  total value of 'Constant alcohol suspension' days
Subjective alcohol craving | At 12, 20 and 32 weeks of stimulation
  change in alcohol urge Visual Analogue Score compared to baseline. ( 0 is no urge, 10 is extreme urge)
Alcohol withdrawal scores | At 12, 20 and 32 weeks of stimulation
  change in Clinical Institute Withdrawal Assessment for Alcohol Scale (CIWA-Ar) score compared to baseline. Minimum score is 0, maximum score is 67, higher the score, alcohol withdrawal is more severe (worse outcome).
Sleep status | At 12, 20 and 32 weeks of stimulation
  Pittsburgh Sleep Quality Index score compared to baseline.
affect status | At 12, 20 and 32 weeks of stimulation
  Hamilton Anxiety Scale-17 and Hamilton Depression Scale score compared to baseline.
Social functionings | At 12, 20 and 32 weeks of stimulation
  Substance Dependence Severity Scale (SDSS) score compared to baseline. Minimum score is 0, maximum score is 20, higher the score, substance dependence is more severe (worse outcome).

OTHER OUTCOMES:
Electrophysiology indicators | Before stimulation and parameter optimization period
  Before stimulation and parameter optimization period, DBS brain electrophysiology study will be conducted, such as electroencephalogram, target Local Field Potential; Observe instant effect to participants at stimulation onset (including instant desire change, emotional change, behavioral change of experimental psychological paradigm and change in brain electrophysiological indicators etc. ), thus to provide evidence for parameter adjustment for the study).
Incidence of adverse events and related data | Collect security data throughout the research period, including AE, SAE, etc.
  1. Adverse events (AE) and device-related adverse events.
  2. Serious adverse events (SAE) and device-related serious adverse events.
  3. Device deficiencies and device malfunctions.
  4. Physical examination and vital signs.
  5. Laboratory check: blood reverse transcription (RT), prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT), Fbg, liver/kidney functions, liver ultrasonic and ECG.
  6. Imaging examination: CT or MRI.
  7. Early drop out ratio due to adverse events.
Positron Emission Topography imaging indicators | Before stimulation and parameter optimization period
  Before DBS implant, use Positron Emission Topography (PET) to study imaging of brain metabolism, receptor and structures. Metabolism features (DA, GABA, Glu) of brain areas including DLPFC, medial prefrontal prefrontal cortex, NAcc, dorsal striatum etc. will be the focus. Patients will be retested for PET after 6 months of implant.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hao, Study Chair — Second Xiangya Hospital of Central South University; Min Zhao, Study Chair — Shanghai Mental Health Center
Locations (4):
- China (4):
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No